CLINICAL TRIAL: NCT05407545
Title: Evaluation of a Motorised Prosthetic Knee
Acronym: MOKI-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Össur Iceland ehf (Industry)
Responsible Party: Principal Investigator, Kevin De Pauw, Prof. Dr., Vrije Universiteit Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EC-2022-184
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Lower Limb Amputation Above Knee (Injury)
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prosthesis (Experimental): A unilateral transfemoral amputee will conduct experiments with the active prosthesis and with the current prosthesis.
  Interventions: Device: Current prosthesis; Device: Active Prosthesis (PowerKnee)

INTERVENTIONS:
Device: Current prosthesis — A unilateral transfemoral amputee will conduct experiments with the current prosthesis
Device: Active Prosthesis (PowerKnee) — A unilateral transfemoral amputee will conduct experiments with the Power Knee. The PowerKnee is an active prosthesis developed by Össur.

SUMMARY:
The study will investigate the effect over time of the Power Knee (Össur) on performance during daily activities in people with a unilateral transfemoral amputation, will determine subjective feelings and gait kinematics over time during daily activities and will investigate the association between subjective feelings and objective outcomes of performing daily activities.

DETAILED DESCRIPTION:
Participants will visit the lab 6 times over a period of 5 weeks. The study includes a familiarisation phase (3 measuring moments) followed by the experimental phase (3 measuring moments). During the measuring sessions, participants will perform four tasks with their current prosthesis and with the Power Knee (Össur). The order in which the devices will be tested, will be reversed on each measuring moment to control for possible order effects and fatigue.

The experimental protocol will entail an L-test and slope walking test that will each be performed 3 times, followed by a 6 minutes of hallway walking (6MWT), 10 min rest and a dual-task 6MWT.

The slope walking test assesses the participants' ability to ascend and descend a 6 m long ramp of 10% inclination as fast as possible. For safety reasons bilateral handrails are warranted. Participants start the test in an upright position in front of the ramp and are asked to ascend the ramp, turn around on the platform, descend the ramp and return to the starting position.

The L-test, requires higher physical activity of the user. During the L-test, participants are asked to rise from a chair, walk 7 meters, turn 90 degrees, walk 3 meters, turn 180 degrees and then return in the same way to the seated position. A total distance of 20 meter is covered.

The 6MWT will be performed on a hallway at a self-selected walking speed, which closely relates to the most efficient walking speed.

The dual-task 6MWT will be compiled out of conducting a 6MWT while performing a cognitive task, i.e. serial subtractions. Serial subtraction is mental arithmetic task that tests attention and working memory. Participants will be asked to continually subtract sevens from a random selected 3-digit number as long as the duration of the test.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transfemoral (above knee) amputation
* Healthy subject
* Medicare Functional Classification Level: K3-4

Exclusion Criteria:

* Any neurological disease
* Upper limb or bilateral amputation
* Stump pain or bad fit of the socket

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Performance | 70 minutes
  Time needed to perform the L-test and slope walking test
Performance | 72 minutes
  Accuracy of the serial subtractions during the dual-6MWT in %
Performance | 144 minutes
  Distance covered during the 6MWT and dual-6MWT

SECONDARY OUTCOMES:
Physiological | 286 minutes
  Heart rate during all tasks in beats per minute
Psychological | 100 minutes
  Visual analogue scale for comfort (score: 0= not comfortable, 100 = comfortable) and fatigue (score: 0= not fatiguing, 100 = fatiguing) during all tasks
Psychological | 96 minutes
  Borg rating of perceived exertion (score: 6 = No exertion at all , 20 = Maximal exertion)
Psychological | 200 minutes
  Perceived workload: Nasa-Task Load Index (score: 0 = minimal workload, 100 = Maximal perceived workload )

CONTACTS AND LOCATIONS:
Overall Officials: Kevin De Pauw, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cox PD, Frengopoulos CA, Hunter SW, Sealy CM, Deathe AB, Payne MWC. Impact of Course Configuration on 6-Minute Walk Test Performance of People with Lower Extremity Amputations. Physiother Can. 2017;69(3):197-203. doi: 10.3138/ptc.2016-24. PMID 30275635
- [Background] Howard CL, Wallace C, Perry B, Stokic DS. Comparison of mobility and user satisfaction between a microprocessor knee and a standard prosthetic knee: a summary of seven single-subject trials. Int J Rehabil Res. 2018 Mar;41(1):63-73. doi: 10.1097/MRR.0000000000000267. PMID 29293160
- [Background] General Assembly of the World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. J Am Coll Dent. 2014 Summer;81(3):14-8. PMID 25951678
- [Background] Gailey RS, Gaunaurd I, Agrawal V, Finnieston A, O'Toole C, Tolchin R. Application of self-report and performance-based outcome measures to determine functional differences between four categories of prosthetic feet. J Rehabil Res Dev. 2012;49(4):597-612. doi: 10.1682/jrrd.2011.04.0077. PMID 22773262
- [Background] Ghillebert J, Bock SD, Flynn L, Geeroms J, Tassignon B, Roelands B, et al. Guidelines and Recommendations to Investigate the Efficacy of a Lower-Limb Prosthetic Device: A Systematic Review. IEEE Transactions on Medical Robotics and Bionics. 2019;1(4):279-96.
- [Background] Williams RM, Turner AP, Orendurff M, Segal AD, Klute GK, Pecoraro J, Czerniecki J. Does having a computerized prosthetic knee influence cognitive performance during amputee walking? Arch Phys Med Rehabil. 2006 Jul;87(7):989-94. doi: 10.1016/j.apmr.2006.03.006. PMID 16813788
- [Background] Omana H, Madou E, Montero-Odasso M, Payne MW, Viana R, Hunter SW. The effect of dual-task testing on the balance and gait of people with lower limb amputations: A systematic review. PM R. 2023 Jan;15(1):94-128. doi: 10.1002/pmrj.12702. Epub 2021 Nov 13. PMID 34464018
- [Background] Morgan SJ, Hafner BJ, Kelly VE. Dual-task walking over a compliant foam surface: A comparison of people with transfemoral amputation and controls. Gait Posture. 2017 Oct;58:41-45. doi: 10.1016/j.gaitpost.2017.07.033. Epub 2017 Jul 10. PMID 28711652
- [Background] Lee KA, Hicks G, Nino-Murcia G. Validity and reliability of a scale to assess fatigue. Psychiatry Res. 1991 Mar;36(3):291-8. doi: 10.1016/0165-1781(91)90027-m. PMID 2062970
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Hart SG, Staveland LE. Development of NASA-TLX (Task Load Index): Results of Empirical and Theoretical Research. In: Hancock PA, Meshkati N, editors. Advances in Psychology. 52: North-Holland; 1988. p. 139-83.
- [Background] De Pauw K, Cherelle P, Tassignon B, Van Cutsem J, Roelands B, Marulanda FG, Lefeber D, Vanderborght B, Meeusen R. Cognitive performance and brain dynamics during walking with a novel bionic foot: A pilot study. PLoS One. 2019 Apr 3;14(4):e0214711. doi: 10.1371/journal.pone.0214711. eCollection 2019. PMID 30943265
- [Derived] Lathouwers E, Maricot A, Tassignon B, Geers S, Flynn L, Verstraten T, De Pauw K. User accommodation to an active microprocessor-controlled knee in individuals with unilateral transfemoral amputation: a 5-week non-randomized trial. J Neuroeng Rehabil. 2025 May 6;22(1):105. doi: 10.1186/s12984-025-01637-5. PMID 40329316